CLINICAL TRIAL: NCT03548727
Title: A Pilot Study to Assess the Feasibility of Pseudo-Simultaneous Imaging of Tumor Hypoxia and Proliferation in Head and Neck Cancer Patients Using PET/CT
Brief Title: Pseudo-Simultaneous Imaging of Tumor Hypoxia and Proliferation in HNC Patients Using PET/CT
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1703018046
Record Dates: First submitted 2018-03-23; First posted 2018-06-07 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: The study includes two arms:
  Arm1: FLT PET/CT on Day1 and Day2 Arm2: Combined FMISO/FLT PET/CT on Day1 and FLT PET/CT on Day2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Repeatability of FLT kinetics (Experimental): Radiotracer: 18F-FLT Dose: 10 mCi Frequency: Two baseline PET/CT at baseline up to 3 days apart.
  Interventions: Diagnostic Test: PET/CT Imaging
- Pseudo-Simultaneous FMISO/FLT PET/CT Imaging (Experimental): Radiotracer: 18F-FLT and 18F-FLT Dose and Frequency: 8 mCi 18F-FLT and 8 mCi 18F-FLT on Day1, the 8mCi 18F-FLT on Day2
  Interventions: Diagnostic Test: PET/CT Imaging

INTERVENTIONS:
Diagnostic Test: PET/CT Imaging — PET/CT Imaging of tumor hypoxia and proliferation

SUMMARY:
66% of HNC patients present with advanced-stage disease at initial diagnosis. The 5-year survival rates for stages IVa, IVb, and IVc are 32%, 25%, and <4% respectively. Accurate pre-treatment staging is vital in determining the optimum procedure for the management of HNC. Early identification of non-responders may allow modification of their treatment through the introduction of more intensive therapies. Identifying prognostic factors that predict patient outcome will ultimately lead to new treatment regimens. Tumor hypoxia and proliferation are two key characteristics of cancer that were shown to correlate with poor response to treatment in HNC. In this proposal, the investigators assess the prognostic values of these two markers. Combining information from these two biological markers shall result in prognostic information superior to those of any of the two separately. Imaging those vital tumor characteristics simultaneously shall provide more coherent assessment of tumor microenvironment than does registration of corresponding images acquired in different imaging session, thus subject to uncertainties resulting from transient biologic changes and image registration process. The investigators propose to use a method that the investigators previously developed to simultaneously and non-invasively image tumor hypoxia (FMISO-PET) and proliferation (FLT-PET) within a single PET/CT study. CT Perfusion scan will be performed 1st, followed by PET imaging with staggered FMISO and FLT injections. FMISO and FLT signals will be separated retrospectively using kinetic modeling. The investigators believe imaging tumor hypoxia and cell proliferation simultaneously yield information underpinning for image-guided and radiobiological based dose painting, adaptive therapy, and patient medical management. If successful, this pilot study will constitute the basis for a NIH grant proposal that aims to improve treatment outcome assessment in HNC.

ELIGIBILITY:
Subject Inclusion Criteria:

* Pathologic Confirmation of HNC
* No prior treatment for this diagnosis of HNC
* Patient to be treated with Radio-Therapy
* Age >= 18 years old
* Karnofsky performance status >= 70%
* Women of childbearing age must have a negative blood pregnancy test.

Exclusion Criteria:

* Women who are pregnant or breast-feeding.
* Severe diabetes (fasting blood glucose > 200- mg/dl)
* Adults who are unable to consent
* Patients who do not agree to share and store data History of lack of tolerance of the standard of care FDG-PET scan previously obtained
* History of previous intolerance of either FMISO or FLT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Simultaneous Imaging of tumor hypoxia and proliferation | 1 year
  To assess the feasibility to tease out the FMISO and FLT kinetics in simultaneous FMISO/FLT PET/CT imaging. FMISO and FLT kinetic parameters will be measured from the combined FMISO/FLT dynamic study. The accuracy of those measurements will be tested by comparing the FLT kinetic measurements deduced from the combined FMISO/FLT study on day1 with those from the sole FLT study of day2.

SECONDARY OUTCOMES:
Repeatability of FLT | 1 year
  To assess the repeatability of FLT kinetics. Subjects will undergo two dynamic FLT PET studies up to 3 days apart. The repeatability of the corresponding kinetic parameters from the two studies will be measured using statistical methods (e.g. Bland-Altman analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Sadek Nehmeh, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Citigroup Biomedical Imaging Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided